CLINICAL TRIAL: NCT00628004
Title: An Open Label Extension Study (to Study DK143WS) Evaluating the Safety and Long-term Safety Follow-up of Biatain Ibu in Painful Chronic Venous Leg Ulcers
Brief Title: Safety Evaluation of Biatain Ibu in Painful Chronic Venous Leg Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DK144WS; DK144WS
Record Dates: First submitted 2008-02-20; First posted 2008-03-04 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Leg Ulcers
MeSH Terms: conditions — Leg Ulcer

STUDY DESIGN:
Masking Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1 (Experimental)
  Interventions: Device: Biatain Ibu
- 2 (Active Comparator)
  Interventions: Device: Local best practice
- No treatment (No Intervention): No treatment as wound was healed

INTERVENTIONS:
Device: Biatain Ibu — Biatain Ibu non-adhesive (Coloplast A/S), a polyurethane foam dressing with an elastic semi-permeable backing film with an added pain relieving medicinal substance ibuprofen (Albermarle Inc.), size 15x15 cm. The product is CE marked.
  Other Names: Coloplast Biatain Ibu
  Arms: 1
Device: Local best practice — N/A - since intervention is "local best practice"
  Arms: 2

SUMMARY:
The objective of this open label extension study (extension to study DK143WS) is to evaluate the safety of Biatain Ibu during 6 -12 weeks of exposure and during a 40 - 46 weeks safety follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* The patient has participated in study DK143WS
* The patient is able to understand the treatment and is willing to comply with the treat-ment regimen.
* The patient is willing and able to give written informed consent

Exclusion Criteria:

* Pregnant or lactating women
* Concomitant participation in other studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2008-05; Primary Completion 2009-07 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Adverse events | Week 1, 6, 20, 33, 46

SECONDARY OUTCOMES:
Clinical occurrences | Week 1, 6, 20, 33, 46
Ulcer area reduction | Week 1, 6, 20, 33, 46
Ulcer status | Week 1, 6, 20, 33, 46
Skin condition at healed ulcer location | Week 1, 6, 20, 33, 46

CONTACTS AND LOCATIONS:
Overall Officials: Karsten Fogh, MD, Principal Investigator — Aarhus University Hospital
Locations (5):
- Denmark (3):
  - Aarhus Universitetshospital, Aarhus
  - Bispebjerg Hospital, Copenhagen
  - Odense Universitets Hospital, Odense
- Georg-August-Universität Göttingen, Göttingen, Germany
- Hospital de Fuenlabrada, Fuenlabrada, Spain